CLINICAL TRIAL: NCT05539430
Title: A Phase 1, Open-Label, Dose Escalation and Expansion, Multicenter Study of Claudin 18.2-Targeted Chimeric Antigen Receptor T-cells in Subjects With Unresectable, Locally Advanced, or Metastatic Gastric, Gastroesophageal Junction (GEJ), Esophageal, or Pancreatic Adenocarcinoma
Brief Title: Claudin 18.2-Targeted Chimeric Antigen Receptor T-cells in Subjects With Unresectable, Locally Advanced, or Metastatic Gastric, Gastroesophageal Junction (GEJ), Esophageal, or Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Legend Biotech USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB1908-1001
Record Dates: First submitted 2022-09-01; First posted 2022-09-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer; Esophageal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental LB1908 (Experimental): Claudin 18.2-Targeted Chimeric Antigen Receptor T-cells
  Interventions: Biological: LB1908

INTERVENTIONS:
Biological: LB1908 — Claudin 18.2-Targeted autologous Chimeric Antigen Receptor T-cells

SUMMARY:
This is a Phase 1, Open-Label, Dose Escalation and Expansion, Multicenter Study of Claudin 18.2-Targeted Chimeric Antigen Receptor T-cells in Subjects with Unresectable, Locally Advanced, or Metastatic Gastric, Gastroesophageal Junction (GEJ), Esophageal, or Pancreatic Adenocarcinoma

DETAILED DESCRIPTION:
This is a Phase 1, open label, dose escalation, multicenter study to evaluate Claudin 18.2-targeting CAR-T cells (LB1908) in adult subjects with unresectable, locally advanced or metastatic gastric, GEJ, esophageal, or pancreatic adenocarcinoma. Patients will be confirmed to have sufficient expression of Claudin 18.2 as part of a prescreening. The study comprises a dose-escalation component (Part A) and a dose-expansion component (Part B). In part A, patients with gastric, GEJ, or esophageal adenocarcinoma will be treated with LB1908 at protocol-defined dose level, with escalation to higher doses in subsequent patients guided by evaluation of protocol-defined dose limiting toxicities (DLTs). Part A will identify the recommended dose for expansion (RDE) to be tested in part B in several cohorts:

* Monotherapy regimen (MR) cohorts: treating second or later line gastric, GEJ, and esophageal adenocarcinoma or pancreatic adenocarcinoma patients as standalone treatment.
* Consolidation regimen (CR) cohorts: treating frontline gastric, GEJ, and esophageal adenocarcinoma or pancreatic adenocarcinoma patients who have achieved disease control with standard of care chemotherapy.

Part B will aim to identify the recommended dose for phase 2 (RP2D)and evaluate preliminary efficacy in these different treatment settings and patient populations.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, all of the following inclusion criteria must be fulfilled.

1. Be willing and able to provide written informed consent.
2. Be a female or male ≥ 18 and ≤ 75 years old at the time of signing of the prescreening ICF.
3. For Part A and Part B Cohort MR1 only:

   1. Subjects with histologically/cytologically confirmed unresectable, locally advanced or metastatic adenocarcinoma of the GC/GEJC/EC for which standard treatment is considered intolerable, unlikely to confer significant clinical benefit, is no longer effective, or subject is ineligible or declines standard therapy.
   2. Subjects must have received prior therapy as follows:

      * Previous treatment must have included a fluoropyrimidine and/or platinum containing regimen. Subjects with HER2-neu-positive (HER2+) disease must have also received prior anti-HER2+ therapy.
      * Neoadjuvant/adjuvant treatment will be considered as a prior regimen if disease progression occurred during treatment or within 6 months of cessation of treatment.

      For Part B Cohort MR2 only:
   3. Subjects with histologically/cytologically confirmed unresectable, locally advanced or metastatic PDAC for which standard treatment is considered intolerable, unlikely to confer significant clinical benefit, is no longer effective, or subject is ineligible or declines standard therapy.
   4. Subjects must have received prior therapy as follows:

      * Previous treatment must have included fluoropyrimidine and/or gemcitabine containing regimen.
      * Neoadjuvant/adjuvant treatment will be considered as a prior regimen if disease progression occurred during treatment or within 6 months of cessation of treatment.

      For Part B Cohort CR1 only:
   5. Subjects with histologically/cytologically confirmed metastatic GC/GEJC/EC with RECIST v1.1 SD or PR at the initial response evaluation during first-line SOC treatment.
   6. Subjects with locally advanced, unresectable disease for whom radiation is not planned may be eligible with Sponsor approval.
   7. Subjects who develop metachronous metastatic disease after prior (neo)adjuvant treatment for previously localized disease are eligible if at least 6 months have elapsed since completion of prior chemotherapy (and disease status is satisfied, as above).
   8. Subjects must be clinically suitable to continue at least part of the initial first-line regimen during LB1908 manufacturing.
   9. Negative for human epidermal growth factor receptor 2 (HER2) or ineligible to receive HER2-directed therapy.
   10. Subjects must have received prior therapy as follows:

       * Acceptable SOC first-line regimens include (but are not limited to) leucovorin/fluorouracil/oxaliplatin (FOLFOX; modifications allowed) and capecitabine/oxaliplatin (CAPOX), with or without an approved immune checkpoint inhibitor.

         * Zolbetuximab is allowable as part of first-line SOC (subjects with prior zolbetuximab exposure require Sponsor approval prior to enrollment)
   11. No investigational therapies in first-line therapy, unless the investigational product is discontinued prior to enrollment on this trial.

       For Part B Cohort CR2 only:
   12. Subjects with metastatic PDAC with RECIST v1.1 SD or PR at the initial response evaluation during first-line SOC treatment.
   13. Subjects with locally advanced, unresectable disease for whom radiation is not planned may be eligible with Sponsor approval.
   14. Subjects who develop metachronous metastatic disease after prior (neo)adjuvant treatment for previously localized disease are eligible if at least 6 months have elapsed since completion of prior chemotherapy (and disease status is satisfied, as above).
   15. Subjects must be clinically suitable to continue at least part of the initial first-line regimen during LB1908 manufacturing.
   16. Subjects must have received prior therapy as follows:

       * Acceptable SOC first-line regimens include (but are not limited to) leucovorin/fluorouracil/irinotecan/oxaliplatin (FOLFIRINOX), nabpaclitaxel/ gemcitabine, and liposomal irinotecan/fluorouracil/leucovorin/oxaliplatin (NALIRIFOX).
       * Prior investigational therapies are exclusionary.
   17. No investigational therapies in first-line therapy, unless the investigational product is discontinued prior to enrollment on this trial.
4. Presence of CLDN18.2 positive tumors with staining intensity of ≥ 1+ in ≥ 50% of tumor cells by immunohistochemistry (IHC) (Performed during Prescreening).

   * Subject has available formalin-fixed, paraffin-embedded (FFPE) tumor specimen in a tissue block or unstained serial slides accompanied by an associated pathology report prior to enrollment. Archival or fresh biopsy tissue is required.
   * If a subject had prior CLDN18.2 targeted therapy, subject may be required to have a formalin-fixed, paraffin-embedded tumor specimen in a tissue block or unstained serial slides accompanied by an associated pathology report that was obtained after exposure to CLDN18.2 targeted therapy, prior to enrollment, and fulfill criteria as outlined (>50% expression) as directed by Sponsor.
5. Presence of ≥ 1 radiologically measurable lesion per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Life expectancy of at least 4 months per Investigator judgment.

Exclusion Criteria:

Subjects are not eligible for this study if they fulfill any of the following exclusion criteria:

1. Prior treatment with cellular immunotherapy (e.g., CAR-T) or gene therapy product.
2. Antitumor therapy prior to Screening as follows (Part A and Part B Monotherapy Regimen [second- or later-line subjects] subjects only):

   * Any systemic anticancer therapy (including investigational) within 7 days or at least 5 halflives, whichever is shorter.
   * Monoclonal antibody therapy within 2 weeks. Type of monoclonal antibody should be communicated with Sponsor.

   Palliative radiotherapy is permitted with a safety break, the length of which is at the discretion of the Investigator. Radiotherapy directed at sites of disease assessment is also permitted at the discretion of the Investigator and exclusion of the radiated site for disease assessments.
3. Unstable/active ulcer, varices, or digestive tract bleeding or recent digestive surgery that may have increased risk of bleeding.
4. Clinically significant ascites, pleural or peritoneal effusions requiring weekly clinical intervention at screening.
5. Subjects who are on therapeutic anticoagulation. (Note: subjects who are on therapeutic antiplatelet therapy or prophylactic anticoagulation are permitted to participate if deemed to not be at an increased risk of bleeding from their underlying disease or procedures and are required to obtain approval from Sponsor. Similarly, subjects who can have therapeutic anticoagulation de-escalated to prophylactic dosing prior to LB1908 infusion are also eligible).
6. Known inherited or acquired immune deficiency without the ability of medical control or normalization.
7. History or known brain metastasis or leptomeningeal metastasis. Part B Cohorts MR1 and MR2: Subjects can have brain metastases if previously treated and confirmed stable for at least 4 weeks prior to study entry.
8. Subjects with heavy tumor burden such as significant lung disease or extensive liver metastases (e.g., > 5 liver lesions or a single dominant lesion > 5 cm in maximal dimension).
9. Active autoimmune disease receiving immunosuppressants (e.g., cyclosporine or high dose systemic steroids) prior to screening as follows:

   * Within 2 weeks or 5 half-lives, whichever is longer (those with inhaled or topical steroids recently or currently are not excluded.)
   * Immune-related AEs due to prior immune checkpoint therapy must be ≤ Grade 1 with no ongoing immunosuppression, including a systemic steroid dose ≤ 20 mg daily of prednisone equivalent.
10. Impaired cardiac function or clinically significant cardiac disease including:

    * Unstable angina or myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to apheresis.
    * New York Heart Association (NYHA) Stage III or IV congestive heart failure.
    * History of medically uncontrolled clinically significant cardiac arrhythmia (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block, or third-degree AV block.
11. Prior or active malignancy other than the study indication requiring active therapy and/or in the judgment of the Investigator or Sponsor may affect the interpretation of the study endpoints, including the following exceptions:

    * Smoldering low grade malignancies may be acceptable as long as the Investigator assesses them of having a significant longer life expectancy than the underlying gastric/pancreatic tumor, after discussion with the Sponsor. Carcinoma in situ.
    * Non-melanoma skin cancer (e.g., basal cell or squamous cell carcinoma).
12. Serious and/or uncontrolled medical condition that, in the Investigator's judgment, would cause unacceptable safety risk, interfere with study procedures or results, or compromise compliance with the protocol, such as:

    * Active, uncontrolled, viral, bacterial, or systemic fungal infection.
    * Requirement of supplemental oxygen to maintain oxygen saturation.
    * Clinical evidence of dementia or altered mental status.
13. Active central nervous system (CNS) disorder, stroke or seizure within 6 months of screening.
14. Current known active infection with human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C virus (HBV/HCV).

    * For subjects who are known carriers of HBV, active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV deoxyribonucleic acid (DNA) viral load per institutional guidelines.
    * For subjects with known history of HCV infection, confirmation of sustained virologic response (SVR) is required for study eligibility, defined as ≥24 weeks from initiation of antiviral therapy.
15. Contraindications or life-threatening allergies, hypersensitivity, or intolerance to LB1908b excipients, such as dimethyl sulfoxide (DMSO); or to fludarabine, cyclophosphamide, or tocilizumab.
16. Ongoing toxicity from previous anticancer therapy that has not resolved to Grade 2 or less, except for alopecia, fatigue, nausea, and constipation.

    For Part B Cohorts CR1 and CR2: toxicity from ongoing chemotherapy that is reversible and expected to resolve (based on the discretion of the treating physician) by the time of LD chemotherapy is not necessarily exclusionary.
17. Any prior ≥ Grade 3 gastritis or gastric mucosal injury with zolbetuximab, or lower grade events that have not recovered to Grade 1 or baseline.
18. Major surgery within 4 weeks prior to enrollment, failure to adequately recover from recent surgery, or planned surgery within 4 weeks after LB1908 administration.
19. Pregnant or breast-feeding.
20. Plans to become pregnant or breastfeed, or father a child within 1 year after receiving a LB1908 infusion.
21. Previous history of allogeneic hematopoietic stem cell transplantation (HSCT), major organ transplant or in preparation for organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of LB1908 and determine the optimal dose or recommended dose for expansion (RDE) | 28 days
  Multiple doses will be tested to establish a recommended dose.
To further characterize the safety and tolerability of LB1908 with the RDE identified in the dose-escalation and determine the recommended Phase 2 dose (RP2D) | 90 days
  Treatment of additional patients at the recommended dose as identified in the initial dose escalation part of the study.

SECONDARY OUTCOMES:
To evaluate the preliminary efficacy of LB1908 | Through study completion, a minimum of 2 years
  Measured by Response Evaluation Criteria In Solid Tumors (RECIST)
To characterize the pharmacokinetics of LB1908 in blood | Through study completion, a minimum of 2 years
  CAR-positive T cell counts, CAR transgene level in blood
To evaluate the immunogenicity of LB1908 | Through study completion, a minimum of 2 years
  Presence of anti-LB1908 antibodies

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - John Theurer Cancer Center at HackensackUMC, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Duke University, Durham, North Carolina
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No